CLINICAL TRIAL: NCT01855529
Title: ROPI Study: Evaluation of the Interest of Ropivacaine Streaming in Postoperative Pain After Mastectomy.
Brief Title: ROPI Study : Ropivacaine Interest in Postsurgical Pain After Mastectomy
Acronym: ROPI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-000227-40
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2016-09

CONDITIONS: Pain After Mastectomy
Keywords: ropivacaine, pain, mastectomy
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine arm (Experimental): Ropivacaïne 2 mg/ml 10ml/h
  Interventions: Drug: Ropivacaine in one arm and placebo (NaCl) in the other arm
- NaCl arm (Placebo Comparator): NaCl 0,9% 250ml 10 ml/h
  Interventions: Drug: Ropivacaine in one arm and placebo (NaCl) in the other arm

INTERVENTIONS:
Drug: Ropivacaine in one arm and placebo (NaCl) in the other arm

SUMMARY:
After surgery for breast cancer, the prevalence of chronic pain is estimated between 20 and 68%. They begin after surgery and may persist until more than 6 months. They respond poorly to opioid analgesics impair the quality of life.

Among the different postoperative analgesic techniques used, the use of a local anesthetic infiltration continues catheter has advantages including improving the quality of analgesia, with a significant decrease in average of VAS (scale visual Analogue), a decrease in morphine consumption, improving the quality of life of patients.

Our study aims to evaluate the effectiveness of a continuous local anesthetic infiltration in the control of postoperative pain after mastectomy.

ELIGIBILITY:
Inclusion Criteria:

Age> 18 years

* ASA I-II, WHO 0-1
* mastectomy alone, mastectomy + GGS + mastectomy CA
* No previous history of chronic pain requiring regular intake of analgesics or long-term
* Failure to take opioids within 30 days before surgery

Exclusion Criteria:

* Long-term treatment analgesic or taking opioids within 30 days before surgery
* Concurrent treatment with a drug test, participation in another therapeutic clinical trial within <30 days
* proven allergy to local anesthetics of the amide
* Skin Inflammation
* Sepsis local
* Kidney failure, liver failure, severe or poorly controlled diabetes
* Inability to respond to the assessment of pain using a visual analogue scale (VAS) or a numerical scale (FR).
* mastectomy with immediate breast reconstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Daily consumption of morphine during the first 48 postoperative hours. | during the first 48 postoperative hours

SECONDARY OUTCOMES:
Determination of Ropivacaine plasma (analytical blank: T0) | T0, the day of surgery
Assessment every 4 hours by the IDE that will support the patient during the first 48 hours, then every analgesic taken: • The intensity of pain, VAS or EN | During the first 48 h after surgery
Assessment every 4 hours by the IDE that will support the patient during the first 48 hours, then every analgesic taken: • The site of pain | during the first 48h after the surgery
Assessment every 4 hours by the IDE that will support the patient during the first 48 hours, then every analgesic taken: A potential analgesics administered | during the first 48h after the surgery
Assessment every 4 hours by the IDE that will support the patient during the first 48 hours, then every analgesic taken: Constant: pulse, blood pressure, tympanic temperature, respiratory rate, sedation (0: awake, 1: sleepy, 2 comatose). | during 48h after the surgery
Assessment every 4 hours by the IDE that will support the patient during the first 48 hours, then every analgesic taken: Possible side effects The most common expected morphine: nausea, vomiting, pruritus, acute urine retention. | during the 48h after the surgery
Assessment every 4 hours by the IDE that will support the patient during the first 48 hours, then every analgesic taken: Possible side effects of ropivacaine expected the most common: nausea, vomiting, headache, dizziness, paresthesias. | during 48 hours after the surgery
Assessment every 4 hours by the IDE that will support the patient during the first 48 hours, then every analgesic taken: Condition of dressing • On any abnormality at the site of administration: local redness, pain, skin warmth, pruritus. | during the 48h after the surgery
Assessment every 4 hours by the IDE that will support the patient during the first 48 hours, then every analgesic taken: Determination of Ropivacaine plasma at T0+ 24 h, T0+48h | during 48h after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France